## {Module Name} Module

## **Brief Substance Craving Scale**

| Agency Name: | Site Name: | |
|---|---|---|
| ID #: | Date:// | |
| | STAFF USE ONLY | |
| A. Identify the primary substance dependence f | Ha<br>Heroin or | or Sedatives (Barbiturates, etc.) 1 Benzos (Valium, Xanax, etc.) 2 Illucinogens (including ecstasy) 3 Alcohol 4 other Opiates (Morphine, etc.) 5 Marijuana 6 nulants (cocaine, amphetamine) 7 |
| Please answer the following questions with re | gard to your craving for the primary drug. | |
| | much I desired this drug in the past 24 hours was | None at all □0 Slight □1 Moderate □2 Considerable □3 Extreme □4 |
| 2. The FREQUENCY of my craving, that is, ho | ow often I desired this drug in the past 24 hours wa | Almost never \( \bigcup_0 \) Almost never \( \bigcup_1 \) Several times \( \bigcup_2 \) Regularly \( \bigcup_3 \) Almost constantly \( \bigcup_4 \) |
| 3. The LENGTH of time I spent in craving this | drug during the past 24 hours was: | None at all □0 Very short □1 Short □2 Somewhat long □3 Very long □4 |
| <b>4.</b> Write in the NUMBER of times you think yo | ou had craving for this drug during the past 24 hor | IIS. |

| ID #: | Date:/ | / |
|---|---|---|
| <b>B.</b> A second craved substance during the past 24 hours <i>Choose only ONE from the following. If NONE, page 15.</i> | | |
| Choose only ONE from the following. If NONE, pl | ease ao noi answer Questions 5-8. | None (STOP) |
| | Downers or Sedati | ives (Barbiturates, etc.) |
| | | s (Valium, Xanax, etc.) $\square$ 2 |
| | | ens (including ecstasy) $\square 3$ |
| | | Alcohol □4 |
| | Heroin or other O | piates (Morphine, etc.) $\square 5$ |
| | | Marijuana 🗖 6 |
| | Stimulants (c | cocaine, amphetamine) $\square$ 7 |
| | Other (specify): | |
| Please answer the following questions with regard to | o a <u>second craved drug</u> . | |
| 5. The INTENSITY of my craving, that is, how much | I desired this drug in the past 24 hours was: | None at all $\Box 0$ |
| | | Slight 🗖 1 |
| | | Moderate □2 |
| | | Considerable $\square$ 3 |
| | | Extreme $\square$ 4 |
| 6. The FREQUENCY of my craving, that is, how often | n I desired this drug in the past 24 hours was: | Never $\square$ 0 |
| | | Almost never $\square$ 1 |
| | | Several times $\square$ 2 |
| | | Regularly $\square$ 3 |
| | | Almost constantly □4 |
| 7. The LENGTH of time I spent in craving this drug de | uring the past 24 hours was: | None at all $\Box 0$ |
| | | Very short □1 |
| | | Short $\square$ 2 |
| | | Somewhat long $\square 3$ |
| | | Very long $\square$ 4 |
| <b>8.</b> Write in the NUMBER of times you think you had o | craving for this drug during the past 24 hours. | |

Reference: Somoza, E., Dyrenforth, S., Goldsmith, J., Mezinskis, J., & Cohen, M., 1995. In search of a universal drug craving scale. Paper presented at the Annual Meeting of the American Psychiatric Association, Miami Florida.